CLINICAL TRIAL: NCT00763217
Title: Characterization of Clinical, Biological and Pharmacological Markers of Stroke Outcome
Brief Title: Clinical Biological and Pharmacological Factors Influencing Stroke Outcome
Acronym: biostroke
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CP 05/15; PHRC 2004/1901 (Other: DHOS)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Stroke
Keywords: inflammation; coagulation; neuroprotection; drugs; clinical neurology; pharmacology; biological factors
MeSH Terms: conditions — Stroke; Inflammation; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stroke patient cohort: Patients with an hemispheric ischemic or hemorrhage stroke hospitalized during the 48h following the beginning of stroke

SUMMARY:
In a previous suty, we have demonstrated that prior transient ischemic attack, treatment lipid-lowering drug or physical activity are associated to a better outcome of stroke. The aim of the study is to understand the mechanisms of this preventive neuroprotection by establishing link between biomarkers and preventive and neuroprotective measures.To answer to the question, we conduct a cohort study of stroke patients.

DETAILED DESCRIPTION:
In the cohort, the severity of stroke (NIHSS) will be correlated with :

* clinical factors,
* pharmacological factors,
* biological factors (inflammatory markers, hemostasis...)

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhage stroke
* hemispheric stroke
* stroke dating from less 48h

Exclusion Criteria:

* non hemispheric stroke
* malformative intracranial hemorrhage
* traumatic intracranial hemorrhage
* subarachnoidal hemorrhage

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of stroke patient
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2005-06; Primary Completion 2009-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
severity of stroke measured by NIH severity score | inclusion, day7, month3, year3

SECONDARY OUTCOMES:
clinical, pharmacological and biological (metabolic, inflammation, hemostasis...) cognitive status | inclusion and year3

CONTACTS AND LOCATIONS:
Overall Officials: regis BORDET, MD,PhD, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital - Service de Neurologie vasculaire, Lille, France

REFERENCES:
- [Derived] Colin O, Labreuche J, Deguil J, Mendyk AM, Deken V, Cordonnier C, Deplanque D, Leys D, Bordet R. Preadmission use of benzodiazepines and stroke outcomes: the Biostroke prospective cohort study. BMJ Open. 2019 Jan 15;9(1):e022720. doi: 10.1136/bmjopen-2018-022720. PMID 30782684
- [Derived] Moulin S, Leys D, Schraen-Maschke S, Bombois S, Mendyk AM, Muhr-Tailleux A, Cordonnier C, Buee L, Pasquier F, Bordet R. Abeta1-40 and Abeta1-42 Plasmatic Levels In Stroke: Influence of Pre-Existing Cognitive Status and Stroke Characteristics. Curr Alzheimer Res. 2017;14(6):686-694. doi: 10.2174/1567205012666151027141730. PMID 26502812